CLINICAL TRIAL: NCT04547595
Title: Assessment of Efficacy of Hypnosis Intervention During Lavage Procedure for Knee Osteoarthrosis
Brief Title: Hypnosis Intervention for the Management of Pain Perception During Joint Lavage
Acronym: HypnoArt
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP200138; 2020-A02333-36 (Other: ID-RCB)
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: hypnosis intervention; analgesics; knee osteoarthritis; joint lavage
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL (No Intervention): Standard care
- Hypnosis (Active Comparator): Standard care + intervention
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — given by Expert in this method
  Other Names: Ericksonienne Method
  Arms: Hypnosis

SUMMARY:
The purpose of this study is to determine whether hypnosis intervention added to usual care is more effective than usual care alone to control pain during lavage procedure in patients with knee osteoarthrosis

DETAILED DESCRIPTION:
Joint lavage can be used in acute knee osteoarthritis, and can be repeated when it is effective. This procedure can generate pain and anxiety which are prevented by systematic prescription of analgesics and anxiolytics. To assess the benefit of hypnosis intervention, the investigators designed a monocentric prospective controlled randomised, single-blind study. Patients with acute and painful knee osteoarthritis, having an indication of lavage according to the rheumatologist, will be randomized to standard care, versus standard care and hypnosis. The hypothesis is that hypnosis intervention will decrease the level of pain during lavage, and the analgesics consumption during the week following the lavage. The sample size will be 100, 50 patients per group. Inclusion is scheduled for 18 months, and duration of the study will be 2 years. The main efficacy criterion is the pain score (assessed using VAS) difference between the 2groups; no interim analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of knee osteoarthritis
* indication for a lavage

Exclusion Criteria:

* People who have had both knees washed on the same day.
* People who have already received a joint lavage.
* Patients with psychotic disorders.
* Refusal to participate.
* People who do not understand and/or speak French or who are deaf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by Visual Analog Scale | One Day, at end of lavage procedure
  VAS range 0-10, 10 for most severe pain

SECONDARY OUTCOMES:
Anxiety assessed by Visual Analog Scale | Day 1, before lavage procedure
  VAS range 0-10, 10 for most severe anxiety
Anxiety assessed by Visual Analog Scale | Day 1, at end of lavage procedure
  VAS range 0-10, 10 for most severe anxiety
Pain assessed by Visual Analog Scale | Day 1, before lavage procedure
  VAS range 0-10, 10 for most severe pain
Pain assessed by Visual Analog Scale | Day 7, after lavage procedure
  VAS range 0-10, 10 for most severe pain -via phone call
Gesture tolerability | Day 1, at end of lavage procedure
  4 points : Perfectly tolerable / tolerable / with difficulty / untolerable
Analgesics consumption | Over 1 week after lavage procedure
  Quantification
Operator Impact | Over 1 week after lavage procedure
  pain VAS by linear regression, adjusted by the 'operator' variable

CONTACTS AND LOCATIONS:
Overall Officials: Anna MOLTO, MD, PhD, Study Chair — APHP
Locations (1):
- Cochin Hospital - Rheumatology department, Paris, France

IPD SHARING:
Plan to Share IPD: No